CLINICAL TRIAL: NCT02055677
Title: Personality Profiles, Values and Empathy: Differences Between Ovo/Lacto-vegetarians and Vegans
Acronym: VegMed 2013
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Universität Duisburg-Essen (Other)
Responsible Party: Principal Investigator, Andreas Michalsen, Prof. Dr. Andreas Michalsen, Charite University, Berlin, Germany
Other Study IDs: VegMed2013
Record Dates: First submitted 2013-10-31; First posted 2014-02-05 (Estimated); Last update posted 2014-07-18 (Estimated); Status verified 2014-07

CONDITIONS: Personality
Keywords: personality profiles; values; empathy; quality of life; vegetarians; vegans

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Main goal is to collect and analyze possible differences between ovo / lacto-vegetarians and vegans with respect to their personality profiles, values and empathy through validated questionnaires. Main hypothesis: vegans and ovo / lacto-vegetarians differ in their personality, empathy and values

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years of age

Exclusion Criteria:

* Age under 18 and above 80 years of age

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 5000-10000 vegetarian volunteers
Sampling Method: Probability Sample
Enrollment: 10000 (Actual)
Dates: Start 2014-01; Primary Completion 2014-04 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Big Five SOEP Inventory | Once at baseline
  Validated Questionnaire

SECONDARY OUTCOMES:
Other Validated Questionnaires | Once at baseline
  WHO Quality of Life Questionnaire Empathizing Scale (Short Form) Portraits Value Questionnaire Likert Scales

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Michalsen, MD, Principal Investigator — Charité Medical University, Germany
Locations (1):
- Charité Medical University, Germany, Berlin, State of Berlin, Germany

REFERENCES:
- [Derived] Kessler CS, Michalsen A, Holler S, Murthy VS, Cramer H. How empathic are vegan medical professionals compared to others? Leads from a paper-pencil-survey. Eur J Clin Nutr. 2018 May;72(5):780-784. doi: 10.1038/s41430-017-0007-8. Epub 2017 Nov 6. PMID 29748650
- See also: Charité Medical University Website — http://www.charite.de